Last updated: March 31, 2023

Mindfulness-based Queer Resilience (MBQR) to Promote Mental and Sexual Health among Sexual and Gender Minority Young Adults: Statistical Analysis Plan

A mixed-methods approach will be used to understand feasibility and acceptability of this randomized controlled trial. Descriptive statistics will be used to summarize feasibility and acceptability measures from the full sample. These measures include recruitment rates, retention/attrition rates, session attendance, Client Satisfaction Questionnaire, and session evaluation form.

In addition, qualitative data from exit interviews will be analyzed using template analysis, a thematic analysis methodology that applies data reduction techniques for rapid turnaround, often used in intervention development and refinement research.